CLINICAL TRIAL: NCT05726500
Title: Evaluation of Regional Ventilation Distribution in Patients Affected by Abdominal Sepsis After Emergent Laparotomy
Acronym: CHESTOMY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Università degli Studi di Ferrara (Other)
Collaborators: University of Milan (Other)
Responsible Party: Principal Investigator, Savino Spadaro, Principal investigator, Università degli Studi di Ferrara
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHESTOMY
Record Dates: First submitted 2023-01-13; First posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Abdominal Sepsis; Acute Respiratory Failure; Ventilation Therapy; Complications; Emergencies
Keywords: Electrical impedance tomography; Emergent laparotomy; Compliance partinioning
MeSH Terms: conditions — Intraabdominal Infections; Emergencies | interventions — Blood Gas Analysis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open Abdomen (Other)
  Interventions: Diagnostic Test: Arterial blood gas analysis; Diagnostic Test: Venous blood gas analysis; Diagnostic Test: Esophageal pressure monitoring; Diagnostic Test: Intrabdominal pressure; Diagnostic Test: Electrical impedance tomopgraphy
- Closed Abdomen (Other)
  Interventions: Diagnostic Test: Arterial blood gas analysis; Diagnostic Test: Venous blood gas analysis; Diagnostic Test: Esophageal pressure monitoring; Diagnostic Test: Intrabdominal pressure; Diagnostic Test: Electrical impedance tomopgraphy

INTERVENTIONS:
Diagnostic Test: Arterial blood gas analysis — The researches will collect 2 ml of arterial blood using an arterial line already in place for clinical purposes to perform and arterial gas analysis.
Diagnostic Test: Venous blood gas analysis — The researches will collect 2 ml of arterial blood using a central venous line already in place for clinical purposes to perform a gas analysis.
Diagnostic Test: Esophageal pressure monitoring — The researchers will position an esophageal balloon to evaluate esophageal pressure
Diagnostic Test: Intrabdominal pressure — The researches will assess intrabdominal pressure using the urinary catheter system already in place for clinical purposes .
Diagnostic Test: Electrical impedance tomopgraphy — The researches will evaluate regional ventilation distribution using Electrical impedance tomography at different levels of positive end-expiratory pressure

SUMMARY:
The goal of this clinical trial is to evaluate regional ventilation distribution in patients admitted to the intensive care unit after emergent laparotomy due to abdominal sepsis. The main question it aims to answer is:

• evaluate if patients admitted after an open abdomen strategy have a different regional ventilation distribution compared to patients in which abdomen is closed at the end of the procedure

Participants will undergo non-invasive monitoring (esophageal pressure and electrical impedance tomography) and an blood gas analysis samples.

Researchers will compare open abdomen group and closed abdomen group to see if the ventilation distribution pattern is different.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 and < 90 years
* Admitted to the ICU after emergent laparotomy for abdominal sepsis
* Acute respiratory failure

Exclusion Criteria:

* Controindications to electrical impedance tomography monitoring
* body mass index > 40 kg/m2
* Haemodinamic instability
* Pneumothorax - Pneumomediastinum
* refusal to participate

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-15 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Chest-wall compliance (Ccw) measured using respiratory parameters from the Ventilator | Day 0
  Different chest wall compliance between the two groups measured using the esophageal catheter. Chest wall compliance will be calculated using the data provided from the respiratory monitoring (i.e. esophageal balloon catheter).
Chest-wall compliance (Ccw) measured using respiratory parameters from the Ventilator | Day 1
  Different chest wall compliance between the two groups measured using the esophageal catheter. Chest wall compliance will be calculated using the data provided from the respiratory monitoring (i.e. esophageal balloon catheter).
Chest-wall compliance (Ccw) measured using respiratory parameters from the Ventilator | Day 2
  Different chest wall compliance between the two groups measured using the esophageal catheter. Chest wall compliance will be calculated using the data provided from the respiratory monitoring (i.e. esophageal balloon catheter).

SECONDARY OUTCOMES:
Regional ventilation distribution measured using Electrical impedance tomography | Day 0
  The researchers will evaluate differences in ventilation distribution pattern among the different weaning trials using Electrical Impedance Tomography and focusing on:
  Regional ventilation distribution Regional inhomogeneity Regional compliance distribution Center of Ventilation Regional ventilation delay Regional compliance
Regional ventilation distribution measured using Electrical impedance tomography | Day 1
  The researchers will evaluate differences in ventilation distribution pattern among the different weaning trials using Electrical Impedance Tomography and focusing on:
  Regional ventilation distribution Regional inhomogeneity Regional compliance distribution Center of Ventilation Regional ventilation delay Regional compliance
Regional ventilation distribution measured using Electrical impedance tomography | Day 2
  The researchers will evaluate differences in ventilation distribution pattern among the different weaning trials using Electrical Impedance Tomography and focusing on:
  Regional ventilation distribution Regional inhomogeneity Regional compliance distribution Center of Ventilation Regional ventilation delay Regional compliance
Mortality in the intensive care unit | Up to 28 days
  Mortality rate in ICU
Infection rate during ICU stay | Up to 28 days
  New diagnosis of infections during the ICU stay

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero Universitaria Sant'Anna, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: No